CLINICAL TRIAL: NCT06218290
Title: A Multicenter, Multidose, Study to Assess the Tolerability and Pharmacokinetics of Oxylanthanum Carbonate at Clinically Effective Doses in Patients With Chronic Kidney Disease on Dialysis
Brief Title: A Study to Assess the Tolerability of Oxylanthanum Carbonate in Patients With Chronic Kidney Disease on Dialysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Unicycive Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UNI-OLC-201
Record Dates: First submitted 2024-01-03; First posted 2024-01-23 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Chronic Kidney Disease Requiring Chronic Dialysis
Keywords: CKD, ESRD
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All Patients (Experimental): All patients with chronic kidney disease with hyperphosphatemia
  Interventions: Drug: Oxylanthanum Carbonate

INTERVENTIONS:
Drug: Oxylanthanum Carbonate — Phosphate Binder to Reduce Hyperphosphatemia
  Other Names: OLC

SUMMARY:
The goal of this clinical study is to test the tolerability of oxylanthanum carbonate (OLC) in patients with chronic kidney disease on hemodialysis and have hyperphosphatemia (too much phosphorus in their blood). The main question it aims to answer is whether patients taking OLC for hyperphosphatemia are able to tolerate the drug.

Participants will continue with their scheduled dialysis treatments and replace their current phosphate binder drug with OLC.

DETAILED DESCRIPTION:
This is a 17-week study consisting of 4 parts. In Part 1, patients are screened for eligibility. In Part 2 patients undergo approximately 3-weeks of washout from previous phosphate binder therapy. Part 3 of the study is up to 6-week titration period where patients are treated with OLC starting at a dose level of 1500 mg/day. At the end of 2 weeks, the dose will be adjusted based on serum phosphate level, up to a maximum dose of 3000 mg/day. Part 4 of the study is a 4-week Maintenance Period with patients treated for 4 weeks on the clinically effective dose of oxylanthanum carbonate (OLC) identified in the Titration Period. Patients will return to the clinic for the End-of-Study Visit on the last day of the 4-week Maintenance Period before restarting their prescribed phosphate binder therapy. The primary endpoint will be to evaluate the tolerability of OLC (as assessed by rate of discontinuations due to treatment-related adverse events) and the secondary endpoints are the evaluation of the safety of clinically effective doses of OLC and evaluate the pharmacokinetics of OLC. Once weekly, at one of the patient's scheduled dialysis appointments and at the End-of-Study Visit, the tolerability will be assessed. After the End-of-Study Visit, patients will reinitiate standard therapy. Toxicity will be assessed during the study based on the severity grade (mild, moderate, or severe) as assessed by the Investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be ≥18 years of age.
2. Patient must be willing and capable of giving written Informed Consent, adhering to dosing and visit schedules, and meeting all study requirements.
3. Patient must be willing and able to swallow whole tablets.
4. Patient has chronic kidney disease and is undergoing, and compliant with, hemodialysis treatment at least 3 times per week for at least 12 weeks prior to signing the ICF, at the Investigator's discretion
5. Patient has mean historical serum phosphorous of ≥4.0 mg/dL and ≤7.0 mg/dL while on a phosphate binder (other than lanthanum carbonate) over the 8 weeks prior to signing the ICF
6. Patient has study specific Screening laboratory serum phosphorus value ≥4.0 mg/dL and ≤7.5 mg/dL during Screening (this value can be repeated up to two times if the value is outside the range).
7. Patient, if on calcimimetic agents or Vitamin D receptor activators (VDRAs), has had no changes in their prescription for at least 4 weeks prior to Day 1 (T1).
8. Patient has a single-pool Kt/V of ≥1.2 during the most recent historical monthly laboratory evaluation.
9. Patient is willing to practice an effective form of contraception from study entry until at least 14 days after the last dose of OLC.
10. Females of childbearing potential must have a negative pregnancy test at Screening.

Exclusion Criteria:

1. Patient with known or suspected intolerance or hypersensitivity to the investigational product or any related lanthanum compound (eg, lanthanum carbonate [Fosrenol]).
2. Patient has had prior treatment with lanthanum-based phosphate binder (eg, lanthanum carbonate [Fosrenol]) within the past 8 weeks prior to signing the ICF.
3. Patient's most recent historical PTH >1500 pg/mL within the last 3 months prior to signing the ICF
4. Patient has received any investigational medicinal product (IMP) in a clinical research study within the 30 days prior to Day 1, or less than 5 elimination half-lives prior to Day 1, whichever is longer.
5. Patient is unable to take drugs orally due to disorders or diseases that may affect gastrointestinal function, such as inflammatory bowel diseases (eg, Crohn's disease, ulcerative colitis) or malabsorption syndrome, or procedures that may affect gastrointestinal function, such as gastrectomy, enterectomy, or colectomy as assessed by the Investigator.
6. Patient has a known history of drug or alcohol abuse that the Investigator assesses would interfere with participation in the study.
7. Patient has an active uncontrolled infection on Day 1 in the opinion of the Investigator
8. Patient has an underlying medical condition or other serious illness that would not be appropriate for this study as assessed by the Investigator.
9. Patient is pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-05-29 (Actual); Study Completion 2024-05-29 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-related AEs leading to study drug discontinuation during the Maintenance Period. | 4 weeks
  Tolerability of clinically effective doses of OLC as assessed by the incidence of treatment-related AEs leading to study drug discontinuation during the Maintenance Period.

SECONDARY OUTCOMES:
Adverse Drug Reactions | up to 10 weeks
  To evaluate the safety of clinically effective doses of OLC
Maximum Plasma Concentration (Cmax) of Lanthanum | up to 10 weeks
  To evaluate the pharmacokinetics (PK) of OLC
Area Under the Concentration-Time Curve (AUC) of Lanthanum | up to 10 weeks
  To evaluate the pharmacokinetics (PK) of OLC
Time to Peak Plasma Concentration (Tmax) of Lanthanum | up to 10 weeks
  To evaluate the pharmacokinetics (PK) of OLC
Elimination Half-Life (t1/2) of Lanthanum | up to 10 weeks
  To evaluate the pharmacokinetics (PK) of OLC
Change from Baseline in Clinical Laboratory Tests | Up to 10 weeks
  Hematology and Biochemistry

OTHER OUTCOMES:
Patient Satisfaction Questionnaire | up to 10 weeks
  Assessment of patient satisfaction with OLC treatment

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - US Renal Care, Pine Bluff, Arkansas
  - US Renal Care, Fort Myers, Florida
  - US Renal Care, Gallup, New Mexico
  - US Renal Care, Cheektowaga, New York
  - US Renal Care, Toledo, Ohio
  - US Renal Care, San Antonio, Texas
  - Clinical Advancement Center, PLLC, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol, CSR
Time Frame: June 2024

REFERENCES:
- [Derived] Block GA, Chertow GM, Reddy G, Hasal SJ, Mourya S, Block M, Gupta S, Pergola PE. A Phase 2 Clinical Trial of Oxylanthanum Carbonate in Patients Receiving Maintenance Hemodialysis with Hyperphosphatemia. Clin J Am Soc Nephrol. 2025 Jul 14;20(9):1259-1267. doi: 10.2215/CJN.0000000780. PMID 40658981
- [Derived] Mathur V, Walker M, Hasal S, Reddy G, Gupta S. Two-Way Randomized Crossover Study to Establish Pharmacodynamic Bioequivalence Between Oxylanthanum Carbonate and Lanthanum Carbonate. Clin Ther. 2025 Jan;47(1):70-75. doi: 10.1016/j.clinthera.2024.11.009. Epub 2024 Nov 30. PMID 39617673